CLINICAL TRIAL: NCT04831866
Title: Coronavirus Disease 2019 (COVID-19) Surveillance and Exposure Testing in School Communities
Brief Title: COVID-19 Surveillance and Exposure Testing in School Communities
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108049
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surveillance Cohort: Surveillance Cohort: Schools participating in this cohort will be performing surveillance testing weekly on approximately 10-20% of students and 100% of staff.
- Exposure Cohort: Exposure Cohort: Schools participating in this cohort will be performing exposure testing on students and staff who have been identified as having close contact with school members diagnosed with SARS-CoV-2 infection.

SUMMARY:
This is a prospective, observational study of COVID-19 surveillance and exposure testing in school communities. Participating school communities are providing severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) tests to students and staff at their schools per school, local, and national guidelines. This study will combine data received from the schools with data collected directly from participants to guide analysis of the co-primary objectives. Participants will be grouped into two different cohorts, depending on each school's SARS-CoV-2 test administration practices.

Surveillance Cohort: Schools participating in this cohort will be performing surveillance testing weekly on approximately 10-20% of students and 100% of staff.

Exposure Cohort: Schools participating in this cohort will be performing exposure testing on students and staff who have been identified as having close contact with school members diagnosed with SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Data from all participating school communities will be included in this study (no inclusion/exclusion criteria will be assessed).

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All students and staff who are members of participating school communities will be given the opportunity to consent to this study. Both children and adult school community members will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Evaluate secondary transmission/prevalence of SARS-CoV-2 in Kindergarten through 12th grade schools in the Surveillance Cohort. | 2 years
  Proportion of students/staff with positive SARS-CoV-2 test identified by surveillance testing.
Evaluate secondary transmission/prevalence of SARS-CoV-2 in Kindergarten through 12th grade schools in the Exposure Cohort. | 2 years
  Proportion of students/staff with positive SARS-CoV-2 test following within-school exposure.
Describe return to school outcomes in Kindergarten through 12th grade schools in Surveillance Cohort. | 2 years
  Proportion of students who return to in-person education in Fall 2021, Spring 2022, and Fall 2022 from participating schools conducting surveillance testing compared to districts without testing.
Describe return to school outcomes in Kindergarten through 12th grade schools in Exposure Cohort. | 2 years
  Mean time to return-to-school after SARS-CoV-2 exposure in the month after initiation of the school-provided testing program compared to the month prior to initiation of the school-provided testing program.

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Durham Charter Schools, Durham, North Carolina
  - Iredell-Statesville Schools, Statesville, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalu IC, Zimmerman KO, Goldman JL, Keener Mast D, Blakemore AM, Moorthy G, Boutzoukas AE, Campbell MM, Uthappa D, DeLaRosa J, Potts JM, Edwards LJ, Selvarangan R, Benjamin DK, Mann TK, Schuster JE. SARS-CoV-2 Screening Testing Programs for Safe In-person Learning in K-12 Schools. J Pediatric Infect Dis Soc. 2023 Feb 27;12(2):64-72. doi: 10.1093/jpids/piac119. PMID 36412278